CLINICAL TRIAL: NCT00004124
Title: Adjuvant Androgen Deprivation Versus Mitoxantrone Plus Prednisone Plus Androgen Deprivation in Selected High-Risk Prostate Cancer Patients Following Radical Prostatectomy
Brief Title: S9921, Hormone Therapy With or Without Mitoxantrone and Prednisone in Patients Who Have Undergone Radical Prostatectomy for Prostate Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: SWOG Cancer Research Network (Network)
Collaborators: National Cancer Institute (NCI) (NIH); Cancer and Leukemia Group B (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000067352; S9921 (Other: SWOG); CALGB-99904 (Other: CALGB); U10CA032102 (NIH)
Record Dates: First submitted 1999-12-10; First posted 2003-01-27 (Estimated); Results first posted 2018-09-04 (Actual); Last update posted 2022-12-30 (Actual); Status verified 2022-12

CONDITIONS: Prostate Cancer
Keywords: adenocarcinoma of the prostate; stage I prostate cancer; stage II prostate cancer; stage III prostate cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — bicalutamide; Goserelin; Mitoxantrone; Prednisone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- bicalutamide, goserelin (Active Comparator): androgen deprivation
  Interventions: Drug: bicalutamide; Drug: goserelin
- bicalutamide, goserelin, mitoxantrone, prednisone (Experimental): androgen deprivation plus mitoxantrone, prednisone
  Interventions: Drug: bicalutamide; Drug: goserelin; Drug: mitoxantrone hydrochloride; Drug: prednisone

INTERVENTIONS:
Drug: bicalutamide
  Other Names: Casodex
Drug: goserelin
  Other Names: Zoladex
Drug: mitoxantrone hydrochloride
  Arms: bicalutamide, goserelin, mitoxantrone, prednisone
Drug: prednisone
  Arms: bicalutamide, goserelin, mitoxantrone, prednisone

SUMMARY:
RATIONALE: Hormones can stimulate the production of prostate cancer cells. Hormone therapy may fight prostate cancer by reducing the production of androgens. Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. It is not yet known whether hormone therapy plus mitoxantrone and prednisone is more effective than hormone therapy alone for prostate cancer.

PURPOSE: This randomized phase III trial is studying hormone therapy, mitoxantrone, and prednisone to see how well they work compared to hormone therapy alone in treating patients who have undergone radical prostatectomy for prostate cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Compare the overall and disease-free survival of patients with high-risk adenocarcinoma of the prostate treated with adjuvant androgen deprivation therapy with or without mitoxantrone and prednisone after radical prostatectomy.
* Compare the qualitative and quantitative toxic effects of these regimens in this patient population.
* Compare the prostate-specific antigen (PSA) progression-free survival rate in patient treated with these regimens.
* Determine whether PSA progression is a surrogate endpoint for survival or disease-free survival in this patient population.

OUTLINE: This is a randomized, multicenter study. Patients are stratified according to surgical extent of disease (organ confined vs not organ confined, but N0 vs N1), Gleason's sum (less than 7 vs 7 vs greater than 7), and planned radiotherapy (yes vs no). Patients are randomized to one of two treatment arms.

* Arm I:Patients receive goserelin subcutaneously once every 13 weeks (8 injections total) and oral bicalutamide once daily for 2 years in the absence of disease progression or unacceptable toxicity.
* Arm II:Patients receive mitoxantrone IV over 30 minutes on day 1 and oral prednisone twice daily on days 1-21. Treatment repeats every 3 weeks for 6 courses in the absence of disease progression or unacceptable toxicity. Patients also receive hormonal therapy as in arm I beginning concurrently with the initiation of mitoxantrone and prednisone.

Patients may undergo radiotherapy 5 days a week for 6.5-7.8 weeks beginning anytime (arm I) or after completion of chemotherapy (arm II), at the discretion of the physician, in the absence of disease progression or unacceptable toxicity.

Patients are offered the possibility to participate in biomarker research by allowing their tissue/blood to be studied.

Patients are followed every 6 months for 2 years and then annually for up to 13 years.

PROJECTED ACCRUAL: A total of 1,360 patients (680 per treatment arm) will be accrued for this study within 9.5 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed stage T1-T3 adenocarcinoma of the prostate before radical prostatectomy and lymph node dissection

  * Must have undergone prostatectomy within the past 120 days
* Must meet at least 1 of the following pathologic criteria:

  * Gleason sum at least 8
  * pT3b (seminal vesicle), pT4, or N1
  * Gleason sum of 7 and positive margin
  * Preoperative PSA greater than 15 ng/mL, Gleason score greater than 7, or PSA level greater than 10 ng/mL and Gleason score greater than 6
* Must have an undetectable PSA (no greater than 0.2 ng/mL) documented after surgery or prior to adjuvant hormonal therapy (for patients initiating adjuvant hormonal therapy prior to study)
* No evidence of metastatic disease on bone scan if PSA is 20 ng/mL or greater at clinical diagnosis
* No distant metastatic disease

PATIENT CHARACTERISTICS:

Performance status:

* SWOG 0-1

Life expectancy:

* Not specified

Hematopoietic:

* Not specified

Hepatic:

* Not specified

Renal:

* Not specified

Cardiovascular:

* No uncontrolled congestive heart failure
* If history of cardiac disease, LVEF at least 50% by MUGA scan or 2-D echocardiogram

Other:

* No HIV positivity
* No other prior malignancy within the past 5 years except adequately treated basal cell or squamous cell skin cancer or stage I or II cancer that is currently in complete remission

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* Not specified

Chemotherapy:

* Not specified

Endocrine therapy:

* Prior neoadjuvant hormonal therapy of no more than 4 months duration before radical prostatectomy allowed
* Other concurrent adjuvant hormonal therapy allowed if initiated prior to study
* Concurrent low-dose megestrol (less than 40 mg/day) for hot flashes allowed

Radiotherapy:

* No prior radiotherapy
* No concurrent whole pelvis irradiation
* Concurrent radiotherapy allowed at the discretion of the physician

Surgery:

* See Disease Characteristics
* See Endocrine therapy
* Recovered from prior surgery

Other:

* No other prior or concurrent therapy for adenocarcinoma of the prostate

Ages: 18 Years to 120 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 983 (Actual)
Dates: Start 1999-10-15 (Actual); Primary Completion 2017-08-12 (Actual); Study Completion 2018-05-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: L. Michael Glode, MD, Study Chair — University of Colorado, Denver; Nancy A. Dawson, MD, Study Chair — University of Maryland Greenebaum Cancer Center
Locations (234):
- United States (234):
  - Alaska Regional Hospital Cancer Center, Anchorage, Alaska
  - Providence Cancer Center, Anchorage, Alaska
  - Banner Thunderbird Medical Center, Glendale, Arizona
  - Banner Good Samaritan Medical Center, Phoenix, Arizona
  - CCOP - Western Regional, Arizona, Phoenix, Arizona
  - Arkansas Cancer Research Center at University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - Highlands Oncology Group - Springdale, Springdale, Arkansas
  - Alta Bates Comprehensive Cancer Center, Berkeley, California
  - Peninsula Medical Center, Burlingame, California
  - California Cancer Care, Incorporated, Greenbrae, California
  - Marin Cancer Institute at Marin General Hospital, Greenbrae, California
  - Sutter Health - Western Division Cancer Research Group, Greenbrae, California
  - Naval Medical Center - San Diego, San Diego, California
  - San Francisco General Hospital Medical Center, San Francisco, California
  - UCSF Comprehensive Cancer Center, San Francisco, California
  - California Pacific Medical Center - California Campus, San Francisco, California
  - Veterans Affairs Medical Center - San Francisco, San Francisco, California
  - Cancer Center of Santa Barbara, Santa Barbara, California
  - Sansum Medical Clinic, Santa Barbara, California
  - Santa Barbara Hematology Oncology Medical Group at Cancer Center of Santa Barbara, Santa Barbara, California
  - Santa Barbara Hematology Oncology - Solvang, Solvang, California
  - Sutter Solano Medical Center, Vallejo, California
  - Memorial Hospital, Colorado Springs, Colorado
  - North Colorado Medical Center, Greeley, Colorado
  - McKee Medical Center, Loveland, Colorado
  - Eastern Connecticut Hematology and Oncology Associates, Norwich, Connecticut
  - Carl and Dorothy Bennett Cancer Center at Stamford Hospital, Stamford, Connecticut
  - Lombardi Comprehensive Cancer Center at Georgetown University Medical Center, Washington D.C., District of Columbia
  - MBCCOP - Medical College of Georgia Cancer Center, Augusta, Georgia
  - Northeast Georgia Medical Center, Gainesville, Georgia
  - Tripler Army Medical Center, Honolulu, Hawaii
  - Saint Anthony's Hospital at Saint Anthony's Health Center, Alton, Illinois
  - Rush-Copley Cancer Care Center, Aurora, Illinois
  - Good Shepherd Hospital, Barrington, Illinois
  - Robert H. Lurie Comprehensive Cancer Center at Northwestern University, Chicago, Illinois
  - Hematology and Oncology Associates, Chicago, Illinois
  - Veterans Affairs Medical Center - Lakeside Chicago, Chicago, Illinois
  - University of Illinois Cancer Center, Chicago, Illinois
  - Veterans Affairs Medical Center - Chicago Westside Hospital, Chicago, Illinois
  - Mercy Hospital and Medical Center, Chicago, Illinois
  - Swedish Covenant Hospital, Chicago, Illinois
  - University of Chicago Cancer Research Center, Chicago, Illinois
  - Creticos Cancer Center at Advocate Illinois Masonic Medical Center, Chicago, Illinois
  - Advocate Good Samaritan Hospital, Downers Grove, Illinois
  - Evanston Northwestern Healthcare - Evanston Hospital, Evanston, Illinois
  - Veterans Affairs Medical Center - Hines, Hines, Illinois
  - Midwest Center for Hematology/Oncology, Joliet, Illinois
  - Joliet Oncology-Hematology Associates, Limited - West, Joliet, Illinois
  - La Grange Memorial Hospital, La Grange, Illinois
  - North Shore Oncology and Hematology Associates, Limited - Libertyville, Libertyville, Illinois
  - Cardinal Bernardin Cancer Center at Loyola University Medical Center, Maywood, Illinois
  - Good Samaritan Regional Health Center, Mount Vernon, Illinois
  - Cancer Care and Hematology Specialists of Chicagoland - Niles, Niles, Illinois
  - Mid-Illinois Hematology-Oncology Associates at Community Cancer Center, Normal, Illinois
  - Cancer Care Center at Advocate Lutheran Hospital, Park Ridge, Illinois
  - Hematology Oncology Associates - Skokie, Skokie, Illinois
  - Hematology/Oncology of the North Shore at Gross Point Medical Center, Skokie, Illinois
  - Carle Cancer Center at Carle Foundation Hospital, Urbana, Illinois
  - CCOP - Carle Cancer Center, Urbana, Illinois
  - Oncology/Hematology Associates of Southwest Indiana at St. Mary's Cancer Center, Evansville, Indiana
  - Indiana University Cancer Center, Indianapolis, Indiana
  - Saint Anthony Memorial Health Centers, Michigan City, Indiana
  - McFarland Clinic, PC, Ames, Iowa
  - St. Luke's Hospital, Cedar Rapids, Iowa
  - Cedar Rapids Oncology Associates, Cedar Rapids, Iowa
  - Mercy Regional Cancer Center at Mercy Medical Center, Cedar Rapids, Iowa
  - Cedar Valley Medical Specialists, PC - West Ridgeway Avenue, Waterloo, Iowa
  - Covenant Cancer Treatment Center, Waterloo, Iowa
  - Cancer Center of Kansas, PA - Chanute, Chanute, Kansas
  - Cancer Center of Kansas, PA - Dodge City, Dodge City, Kansas
  - Cancer Center of Kansas, PA - El Dorado, El Dorado, Kansas
  - Veterans Affairs Medical Center - Kansas City, Kansas City, Kansas
  - Cancer Center of Kansas, PA - Kingman, Kingman, Kansas
  - Southwest Medical Center, Liberal, Kansas
  - Cancer Center of Kansas, PA - Newton, Newton, Kansas
  - Cancer Center of Kansas, PA - Parsons, Parsons, Kansas
  - Cancer Center of Kansas, PA - Pratt, Pratt, Kansas
  - Cancer Center of Kansas, PA - Salina, Salina, Kansas
  - Cancer Center of Kansas, PA - Wellington, Wellington, Kansas
  - Associates in Womens Health, PA - North Review, Wichita, Kansas
  - Cancer Center of Kansas, PA - Medical Arts Tower, Wichita, Kansas
  - Cancer Center of Kansas, PA - Wichita, Wichita, Kansas
  - CCOP - Wichita, Wichita, Kansas
  - Via Christi Cancer Center at Via Christi Regional Medical Center, Wichita, Kansas
  - Wesley Medical Center, Wichita, Kansas
  - Cancer Center of Kansas, PA - Winfield, Winfield, Kansas
  - Markey Cancer Center at University of Kentucky Chandler Medical Center, Lexington, Kentucky
  - Louisiana State University Health Sciences Center - Monroe, Monroe, Louisiana
  - Veterans Affairs Medical Center - Shreveport, Shreveport, Louisiana
  - Feist-Weiller Cancer Center at Louisiana State University Health Sciences, Shreveport, Louisiana
  - Cancer Research Center at Boston Medical Center, Boston, Massachusetts
  - Lahey Clinic Medical Center - Burlington, Burlington, Massachusetts
  - Commonwealth Hematology-Oncology P.C. - Worcester, Worcester, Massachusetts
  - Saint Joseph Mercy Cancer Center, Ann Arbor, Michigan
  - CCOP - Michigan Cancer Research Consortium, Ann Arbor, Michigan
  - University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan
  - Mecosta County Medical Center, Big Rapids, Michigan
  - Barbara Ann Karmanos Cancer Institute, Detroit, Michigan
  - Green Bay Oncology, Limited - Escanaba, Escanaba, Michigan
  - Genesys Hurley Cancer Institute, Flint, Michigan
  - Hurley Medical Center, Flint, Michigan
  - CCOP - Grand Rapids, Grand Rapids, Michigan
  - Lacks Cancer Center at Saint Mary's Health Care, Grand Rapids, Michigan
  - Spectrum Health Hospital - Butterworth Campus, Grand Rapids, Michigan
  - Metro Health Hospital, Grand Rapids, Michigan
  - Van Elslander Cancer Center at St. John Hospital and Medical Center, Grosse Pointe Woods, Michigan
  - Holland Community Hospital, Holland, Michigan
  - Green Bay Oncology, Limited - Iron Mountain, Iron Mountain, Michigan
  - Foote Hospital, Jackson, Michigan
  - Sparrow Regional Cancer Center, Lansing, Michigan
  - Hackley Hospital, Muskegon, Michigan
  - Northern Michigan Hospital, Petoskey, Michigan
  - Mercy Regional Cancer Center at Mercy Hospital, Port Huron, Michigan
  - William Beaumont Hospital - Royal Oak Campus, Royal Oak, Michigan
  - Seton Cancer Institute - Saginaw, Saginaw, Michigan
  - Munson Medical Center, Traverse City, Michigan
  - St. John Macomb Hospital, Warren, Michigan
  - Alexandria, Minnesota
  - Brainerd Medical Center, Brainerd, Minnesota
  - St. Joseph's Medical Center, Brainerd, Minnesota
  - Fergus Falls, Minnesota
  - Chippewa County - Montevideo Hospital, Montevideo, Minnesota
  - CentraCare Clinic - River Campus, Saint Cloud, Minnesota
  - Coborn Cancer Center, Saint Cloud, Minnesota
  - Adult and Pediatric Urology, P.L.L.P., Sartell, Minnesota
  - Saint Francis Medical Center, Cape Girardeau, Missouri
  - Southeast Missouri Regional Cancer Center at Southeast Missouri Hospital, Cape Girardeau, Missouri
  - Saint Luke's Hospital, Chesterfield, Missouri
  - CCOP - Kansas City, Kansas City, Missouri
  - Siteman Cancer Center at Barnes-Jewish Hospital, St Louis, Missouri
  - Missouri Baptist Cancer Center, St Louis, Missouri
  - Arch Medical Services, Incorporated at Center for Cancer Care Research, St Louis, Missouri
  - CCOP - St. Louis-Cape Girardeau, St Louis, Missouri
  - David C. Pratt Cancer Center at St. John's Mercy, St Louis, Missouri
  - CCOP - Montana Cancer Consortium, Billings, Montana
  - Hematology-Oncology Centers of the Northern Rockies - Billings, Billings, Montana
  - St. Vincent Healthcare, Billings, Montana
  - Billings Clinic Cancer Center, Billings, Montana
  - Deaconess Billings Clinic - Downtown, Billings, Montana
  - Bozeman Deaconess Hospital, Bozeman, Montana
  - St. James Community Hospital, Butte, Montana
  - Great Falls Clinic, Great Falls, Montana
  - Sletten Regional Cancer Institute at Benefis Healthcare, Great Falls, Montana
  - Great Falls, Montana
  - St. Peter's Hospital, Helena, Montana
  - Glacier Oncology, PLLC, Kalispell, Montana
  - Kalispell Medical Oncology, Kalispell, Montana
  - Kalispell Regional Medical Center, Kalispell, Montana
  - Community Medical Center, Missoula, Montana
  - Guardian Oncology and Center for Wellness, Missoula, Montana
  - Montana Cancer Specialists at Montana Cancer Center, Missoula, Montana
  - Montana Cancer Center at St. Patrick Hospital and Health Sciences Center, Missoula, Montana
  - Good Samaritan Cancer Center at Good Samaritan Hospital, Kearney, Nebraska
  - University Medical Center of Southern Nevada, Las Vegas, Nevada
  - CCOP - Nevada Cancer Research Foundation, Las Vegas, Nevada
  - Kingsbury Center for Cancer Care at Cheshire Medical Center, Keene, New Hampshire
  - Lakes Region General Hospital, Laconia, New Hampshire
  - Norris Cotton Cancer Center at Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire
  - Elliot Regional Cancer Center at Elliot Hospital, Manchester, New Hampshire
  - Frisbie Memorial Hospital, Rochester, New Hampshire
  - Cancer Institute of New Jersey at Hamilton, Hamilton, New Jersey
  - Mountainside Hospital Cancer Center, Montclair, New Jersey
  - Carol G. Simon Cancer Center at Morristown Memorial Hospital, Morristown, New Jersey
  - Cancer Institute of New Jersey at UMDNJ - Robert Wood Johnson Medical School, New Brunswick, New Jersey
  - University of New Mexico Cancer Research and Treatment Center, Albuquerque, New Mexico
  - Veterans Affairs Medical Center - Brooklyn, Brooklyn, New York
  - Veterans Affairs Medical Center - Buffalo, Buffalo, New York
  - James P. Wilmot Cancer Center at University of Rochester Medical Center, Rochester, New York
  - Duke Comprehensive Cancer Center, Durham, North Carolina
  - Wayne Memorial Hospital, Incorporated, Goldsboro, North Carolina
  - Pardee Memorial Hospital, Hendersonville, North Carolina
  - Lenoir Memorial Cancer Center, Kinston, North Carolina
  - Rutherford Hospital, Rutherfordton, North Carolina
  - Bismarck Cancer Center, Bismarck, North Dakota
  - Cancer Care Center at Medcenter One Hospital, Bismarck, North Dakota
  - Mid Dakota Clinic, PC, Bismarck, North Dakota
  - St. Alexius Medical Center, Bismarck, North Dakota
  - Akron City Hospital, Akron, Ohio
  - Community Hospitals and Wellness Centers - Bryan, Bryan, Ohio
  - Cleveland Clinic Taussig Cancer Center, Cleveland, Ohio
  - Community Oncology Group at Cleveland Clinic Cancer Center, Independence, Ohio
  - St. Rita's Medical Center, Lima, Ohio
  - Cleveland Clinic - Wooster, Wooster, Ohio
  - Tod Children's Hospital - Forum Health, Youngstown, Ohio
  - OU Cancer Institute, Oklahoma City, Oklahoma
  - St. Charles Medical Center - Bend, Bend, Oregon
  - Legacy Mount Hood Medical Center, Gresham, Oregon
  - Providence Milwaukie Hospital, Milwaukie, Oregon
  - Legacy Good Samaritan Hospital & Medical Center Comprehensive Cancer Center, Portland, Oregon
  - Providence Cancer Center at Providence Portland Medical Center, Portland, Oregon
  - CCOP - Columbia River Oncology Program, Portland, Oregon
  - Providence St. Vincent Medical Center, Portland, Oregon
  - Legacy Emanuel Hospital and Health Center & Children's Hospital, Portland, Oregon
  - Legacy Meridian Park Hospital, Tualatin, Oregon
  - Morgan Cancer Center at Lehigh Valley Hospital - Cedar Crest, Allentown, Pennsylvania
  - PinnacleHealth Regional Cancer Center at Polyclinic Hospital, Harrisburg, Pennsylvania
  - Hillman Cancer Center at University of Pittsburgh Cancer Institute, Pittsburgh, Pennsylvania
  - Cancer Care Institute of Carolina at Aiken Regional Medical Centers, Aiken, South Carolina
  - AnMed Health Cancer Center, Anderson, South Carolina
  - Roper St. Francis Cancer Center at Roper Hospital, Charleston, South Carolina
  - Hollings Cancer Center at Medical University of South Carolina, Charleston, South Carolina
  - CCOP - Upstate Carolina, Spartanburg, South Carolina
  - Gibbs Regional Cancer Center at Spartanburg Regional Medical Center, Spartanburg, South Carolina
  - Mountainview Medical, Berlin Corners, Vermont
  - Fletcher Allen Health Care - University Health Center Campus, Burlington, Vermont
  - St. Joseph Cancer Center, Bellingham, Washington
  - Olympic Hematology and Oncology, Bremerton, Washington
  - Skagit Valley Hospital Cancer Care Center, Mount Vernon, Washington
  - Fred Hutchinson Cancer Research Center, Seattle, Washington
  - Harborview Medical Center, Seattle, Washington
  - Minor and James Medical, PLLC, Seattle, Washington
  - Group Health Central Hospital, Seattle, Washington
  - Swedish Cancer Institute at Swedish Medical Center - First Hill Campus, Seattle, Washington
  - Polyclinic First Hill, Seattle, Washington
  - University Cancer Center at University of Washington Medical Center, Seattle, Washington
  - North Puget Oncology at United General Hospital, Sedro-Woolley, Washington
  - Cancer Care Northwest - Spokane South, Spokane, Washington
  - Rockwood Clinic Cancer Treatment Center, Spokane, Washington
  - Madigan Army Medical Center - Tacoma, Tacoma, Washington
  - Southwest Washington Medical Center Cancer Center, Vancouver, Washington
  - Wenatchee Valley Medical Center, Wenatchee, Washington
  - North Star Lodge Cancer Center at Yakima Valley Memorial Hospital, Yakima, Washington
  - Fox Valley Hematology and Oncology - East Grant Street, Appleton, Wisconsin
  - Green Bay Oncology, Limited at St. Vincent Hospital, Green Bay, Wisconsin
  - Green Bay Oncology, Limited at St. Mary's Hospital, Green Bay, Wisconsin
  - St. Mary's Hospital Medical Center - Green Bay, Green Bay, Wisconsin
  - St. Vincent Hospital Regional Cancer Center, Green Bay, Wisconsin
  - Dean Medical Center - Madison, Madison, Wisconsin
  - University of Wisconsin Comprehensive Cancer Center, Madison, Wisconsin
  - Bay Area Cancer Care Center at Bay Area Medical Center, Marinette, Wisconsin
  - Green Bay Oncology, Limited - Oconto Falls, Oconto Falls, Wisconsin
  - Green Bay Oncology, Limited - Sturgeon Bay, Sturgeon Bay, Wisconsin
  - University of Wisconcin Cancer Center at Aspirus Wausau Hospital, Wausau, Wisconsin
  - Welch Cancer Center at Sheridan Memorial Hospital, Sheridan, Wyoming

REFERENCES:
- [Result] Glode LM, Tangen CM, Hussain MH, et al.: Southwest Oncology Group S9921: prolonged event-free survival in high-risk prostate cancer (PC) patients receiving adjuvant androgen deprivation. [Abstract] J Clin Oncol 27 (Suppl 15): A-5009, 2009.
- [Result] Flaig TW, Tangen CM, Hussain MH, Stadler WM, Raghavan D, Crawford ED, Glode LM; Southwest Oncology Group. Randomization reveals unexpected acute leukemias in Southwest Oncology Group prostate cancer trial. J Clin Oncol. 2008 Mar 20;26(9):1532-6. doi: 10.1200/JCO.2007.13.4197. PMID 18349405
- [Result] Glode LM, Hussain MH, Benson MC, et al.: SWOG 9921: a phase III multi-institutional trial of adjuvant therapy for high risk prostate cancer after radical prostatectomy. [Abstract] American Society of Clinical Oncology 2007 Prostate Cancer Symposium, 22-24 February 2007, Orlando, FL. A-349, 2007.
- [Derived] Hussain M, Tangen CM, Thompson IM Jr, Swanson GP, Wood DP, Sakr W, Dawson NA, Haas NB, Flaig TW, Dorff TB, Lin DW, Crawford ED, Quinn DI, Vogelzang NJ, Glode LM. Phase III Intergroup Trial of Adjuvant Androgen Deprivation With or Without Mitoxantrone Plus Prednisone in Patients With High-Risk Prostate Cancer After Radical Prostatectomy: SWOG S9921. J Clin Oncol. 2018 May 20;36(15):1498-1504. doi: 10.1200/JCO.2017.76.4126. Epub 2018 Apr 6. PMID 29624463
- [Derived] Dorff TB, Flaig TW, Tangen CM, Hussain MH, Swanson GP, Wood DP Jr, Sakr WA, Dawson NA, Haas NB, Crawford ED, Vogelzang NJ, Thompson IM, Glode LM. Adjuvant androgen deprivation for high-risk prostate cancer after radical prostatectomy: SWOG S9921 study. J Clin Oncol. 2011 May 20;29(15):2040-5. doi: 10.1200/JCO.2010.32.2776. Epub 2011 Apr 18. PMID 21502546
- See also: SWOG Cancer Research Network website — https://www.swog.org/
- Available data/document: Individual Participant Data Set — https://nctn-data-archive.nci.nih.gov/ — Data Available: Select individual patient-level data from this trial can be requested from the NCTN/NCORP Data Archive.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 983 patients consented and were enrolled to the trial. 22 patients were found to be ineligible per eligibility criteria, and were thus excluded from final analysis.
Groups:
- Arm I: Bicalutamide + Goserelin: Patients receive goserelin subcutaneously once every 13 weeks (8 injections total) and oral bicalutamide once daily for 2 years in the absence of disease progression or unacceptable toxicity.
- Arm II: Mitoxantrone + Prednisone + Bivalutamid + Goserelin: Patients receive mitoxantrone IV over 30 minutes on day 1 and oral prednisone twice daily on days 1-21. Treatment repeats every 3 weeks for 6 courses in the absence of disease progression or unacceptable toxicity. Patients also receive hormonal therapy as in arm I beginning concurrently with the initiation of mitoxantrone and prednisone.
Period: Overall Study
Arm/Group | Arm I: Bicalutamide + Goserelin | Arm II: Mitoxantrone + Prednisone + Bivalutamid + Goserelin
Started (Eligible Patients Enrolled & Randomized to Study) | 481 | 480
Completed (Received Any Protocol Treatment -- population assessable for adverse events.) | 469 | 460
Not Completed | 12 | 20
Not completed — Received no protocol therapy | 12 | 20

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm I: Bicalutamide + Goserelin | Arm II: Mitoxantrone + Prednisone + Bivalutamid + Goserelin | Total
Number analyzed (Participants) | 481 | 480 | 961
Age, Continuous [Median (Full Range); unit: years] | 60 [40 to 82] | 60 [40 to 86] | 60 [40 to 86]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 481 | 480 | 961
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race/Ethnicity: White | 399 | 411 | 810
  Race/Ethnicity: Black | 66 | 50 | 116
  Race/Ethnicity: Asian | 6 | 11 | 17
  Race/Ethnicity: Other | 10 | 8 | 18
PSA at Prostatectomy [Median (Inter-Quartile Range); unit: ng/mL] | 7.9 [5.1 to 12.3] | 7.4 [5.1 to 12.7] | 7.7 [5.1 to 12.5]
Hispanic [Count of Participants; unit: Participants] | 25 | 30 | 55
Disease Extent [Count of Participants; unit: Participants] — Disease Staging Criteria from the Manual for Staging of Cancer, AJCC, Fifth Edition
  Regional Lymph Nodes (N) N0 - No regional lymph node metastasis N1 - Metastasis in a single lymph node or nodes.
  Primary Tumor, Clinical (T) T3 - Tumor extends through the prostatic capsule. Note: Invasion of disease into the prostatic apex or into (but not beyond) the prostatic capsule is not classified as T3 but as T2.
  Participants
    N1 | 79 | 83 | 162
    >= T3 but N0 | 293 | 306 | 599
    Organ Confined | 109 | 91 | 200
Positive Margins from Prostatectomy [Count of Participants; unit: Participants] | 316 | 293 | 609
Intent to Receive Adjuvant RT [Count of Participants; unit: Participants] | 130 | 127 | 257
Gleason Score [Count of Participants; unit: Participants] — This is a 2 to 10 grading system for prostate carcinoma devised by Dr. Donald Gleason in 1977 as a method for predicting the behavior of prostate cancer. Tumors with a low Gleason score are less likely to show aggressive behavior and therefore are less likely to have spread outside of the gland to lymph nodes. To obtain a Gleason score, the dominant tumor pattern is added to the second most prevalent pattern to obtain a number between 2 and 10. If a tumor has patterns 3 and 2, the score would be 5. If the tumor has only one pattern, then the single pattern is added to itself (e.g. 3+3=6).
  Participants
    <= 6 | 10 | 12 | 22
    7 | 215 | 220 | 435
    8 - 10 | 256 | 248 | 504
Risk Groups [Count of Participants; unit: Participants] — Node Positive-- Prostate Cancer with metastases to lymph nodes
  pT3b - The pathological grade of the primary tumor where the tumor presents with extraprostatic extension with seminal vesicle invasion. Defined by the Manual for Staging of Cancer, AJCC, Fifth Edition.
  Positive Margins -- cancer cells detected on edge of tissue removed from patient during radical prostatectomy.
  PSA -- Prostate Specific Antigen -- a blood test that used to screen for cancer of the prostate and to monitor treatment of the disease.
  Participants
    Node Positive | 79 | 83 | 162
    Gleason Score >= 8 or pT3b | 276 | 296 | 572
    Gleason Score<8 w/Positive Margins or PSA>10 ng/mL | 126 | 101 | 227

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival
Description: Measured from date of randomization to date of death from any cause. Patient known to be alive are censored at date of last contact.
Time Frame: at 10 Years
Measure: Number; unit: percentage of probability of survival
Arm/Group | Arm I: Bicalutamide + Goserelin | Arm II: Mitoxantrone + Prednisone + Bivalutamid + Goserelin
Number analyzed (Participants) | 481 | 480
percentage of probability of survival | 87 | 86
Statistical Analysis 1: Comparison: Arm I: Bicalutamide + Goserelin vs Arm II: Mitoxantrone + Prednisone + Bivalutamid + Goserelin; Test type: Superiority; p = 0.70, Regression, Cox; Hazard Ratio (HR) = 1.06, 95% CI 2-sided [0.79 to 1.43]

2. Primary Outcome: Disease Free Survival
Description: Measured from date of randomization to date of first observation of recurrence or death due to any cause. Patients without recurrence are censored at date of last contact.
Time Frame: at 10 Years
Population: Intent-to-treat
Measure: Number; unit: percentage of probability of survival
Arm/Group | Arm I: Bicalutamide + Goserelin | Arm II: Mitoxantrone + Prednisone + Bivalutamid + Goserelin
Number analyzed (Participants) | 480 | 481
percentage of probability of survival | 72 | 72
Statistical Analysis 1: Comparison: Arm I: Bicalutamide + Goserelin vs Arm II: Mitoxantrone + Prednisone + Bivalutamid + Goserelin; Test type: Superiority; p = 0.94, Regression, Cox; Hazard Ratio (HR) = 1.01, 95% CI 2-sided [0.80 to 1.27]

3. Secondary Outcome: Compare Qualitative and Quantitative Toxicities of These Regimens in These Patients
Description: Number of patients with adverse events that are related to study drug
Time Frame: Up to 22 months from registration
Population: All eligible patients who received protocol therapy
Measure: Number; unit: Participants
Arm/Group | Arm I: Bicalutamide + Goserelin | Arm II: Mitoxantrone + Prednisone + Bivalutamid + Goserelin
Number analyzed (Participants) | 469 | 460
Participants
  Abdominal pain/cramping | 19 | 41
  Abscess | 0 | 1
  Alkaline phosphatase increase | 11 | 11
  Allergic reaction | 1 | 5
  Allergic rhinitis | 2 | 16
  Alopecia | 91 | 131
  Anal incontinence | 2 | 2
  Anemia | 52 | 141
  Anorexia | 7 | 41
  Anxiety/agitation | 52 | 62
  Apnea | 1 | 1
  Arrhythmia, NOS | 0 | 1
  Arthralgia | 43 | 64
  Arthritis | 17 | 17
  Ataxia (incoordination) | 1 | 1
  Bilirubin increase | 5 | 20
  Blurred vision | 3 | 6
  Bone pain | 19 | 34
  Bruising | 1 | 14
  CPK increase | 0 | 2
  Cardiac ischemia/infarction | 1 | 1
  Cardiovascular-other | 0 | 5
  Cataract | 5 | 6
  Cerebrovascular ischemia | 1 | 0
  Chest pain,not cardio or pleur | 11 | 19
  Conduction abnormality/block | 1 | 0
  Confusion | 6 | 14
  Conjunctivitis | 0 | 4
  Constipation/bowel obstruction | 57 | 117
  Cough | 10 | 34
  Creatinine increase | 7 | 17
  Cushingoid appearance | 0 | 8
  Dehydration | 0 | 6
  Depression | 80 | 85
  Diarrhea without colostomy | 55 | 75
  Dizziness/light headedness | 33 | 71
  Dry eye | 1 | 5
  Dry skin | 11 | 28
  Dysmenorrhea | 0 | 1
  Dyspepsia/heartburn | 7 | 44
  Dyspnea | 21 | 49
  Dysuria | 14 | 11
  Ear-other | 0 | 2
  Edema | 40 | 56
  Endocrine-other | 3 | 2
  Epistaxis | 0 | 2
  Erectile impotence | 181 | 146
  Eryth/rash/eruption/desq, NOS | 0 | 2
  Esophagitis/dysphagia | 2 | 13
  Eye-other | 1 | 6
  Fatigue/malaise/lethargy | 258 | 357
  Febrile neutropenia | 0 | 2
  Feminization of male | 1 | 0
  Fever without neutropenia | 0 | 9
  Fever, NOS | 1 | 6
  Flatulence | 2 | 3
  Flu-like symptoms-other | 2 | 6
  Flushing | 5 | 4
  GGT increase | 1 | 0
  GI Mucositis, NOS | 0 | 10
  GI-other | 12 | 20
  GU-other | 9 | 9
  Gastritis | 2 | 0
  Gastritis/ulcer, NOS | 0 | 1
  Glaucoma | 2 | 0
  Gynecomastia | 140 | 100
  Headache | 37 | 82
  Hematologic-other | 1 | 1
  Hematuria | 9 | 13
  Hemolysis | 0 | 1
  Hemoptysis | 0 | 1
  Hemorrhage-other | 1 | 4
  Hiccoughs | 0 | 4
  Hot flashes | 439 | 422
  Hypercalcemia | 4 | 5
  Hypercholesterolemia | 5 | 2
  Hyperglycemia | 44 | 78
  Hyperkalemia | 0 | 4
  Hypermagnesemia | 0 | 1
  Hypernatremia | 0 | 4
  Hypertension | 38 | 38
  Hypertriglyceridemia | 2 | 0
  Hypoalbuminemia | 1 | 6
  Hypocalcemia | 1 | 7
  Hypoglycemia | 0 | 1
  Hypokalemia | 8 | 11
  Hypomagnesemia | 1 | 1
  Hyponatremia | 3 | 2
  Hypotension | 3 | 11
  Hypothyroidism | 2 | 0
  Hypoxia | 0 | 4
  Incontinence | 88 | 71
  Infection w/o 3-4 neutropenia | 5 | 10
  Infection with 3-4 neutropenia | 0 | 2
  Infection, unk ANC | 1 | 4
  Inner ear-hearing loss | 3 | 2
  Insomnia | 79 | 92
  Invol. movement/restlessness | 2 | 2
  Joint,muscle,bone-other | 11 | 27
  LVEF decrease/CHF | 0 | 8
  Leukopenia | 14 | 317
  Libido loss | 163 | 133
  Local injection site reaction | 11 | 17
  Lung-other | 0 | 2
  Lymphopenia | 4 | 49
  Male infertility | 2 | 3
  Melena/ GI bleeding | 0 | 2
  Memory loss | 15 | 12
  Metabolic-other | 0 | 1
  Middle ear-hearing loss/otitis | 0 | 1
  Mood/consciousness change, NOS | 2 | 3
  Mouth dryness | 10 | 13
  Muscle weakness (not neuro) | 55 | 77
  Myalgia | 26 | 45
  Myalgia/arthralgia, NOS | 1 | 12
  Myocarditis | 0 | 1
  Nail changes | 4 | 57
  Nausea | 26 | 205
  Neuro-other | 5 | 4
  Neuropathic pain | 0 | 1
  Neutropenia/granulocytopenia | 11 | 239
  PRBC transfusion | 0 | 3
  Pain-other | 112 | 127
  Palpitations | 1 | 6
  Pelvic pain | 9 | 11
  Pericar. effusion/pericarditis | 0 | 1
  Personality/behavioral change | 12 | 11
  Phlebitis | 0 | 5
  Pigmentation changes/yellowing | 0 | 3
  Pleural effusions | 0 | 1
  Pneumonitis/infiltrates | 0 | 1
  Proctitis | 4 | 4
  Proteinuria | 3 | 1
  Pruritus | 13 | 23
  RT-GI mucositis, NOS | 0 | 1
  RT-focal dermatitis, NOS | 3 | 1
  RT-late bladder morbidity | 1 | 0
  RT-late intestinal morbidity | 2 | 1
  RT-pain | 1 | 0
  Rash/desquamation | 46 | 63
  Rectal bleeding/hematochezia | 12 | 10
  Rectal/perirectal pain | 7 | 5
  Respiratory infect w/o neutrop | 1 | 7
  Respiratory infection, unk ANC | 1 | 8
  Rigors/chills | 7 | 24
  SGOT (AST) increase | 42 | 42
  SGPT (ALT) increase | 22 | 26
  Salivary change, NOS | 0 | 1
  Second primary | 0 | 6
  Seizures | 1 | 1
  Sensory neuropathy | 37 | 57
  Sexual/reproductive-other | 2 | 1
  Sinus bradycardia | 0 | 4
  Skin-other | 11 | 11
  Speech impairment | 0 | 1
  Stomatitis/pharyngitis | 5 | 49
  Supraventricular arrhythmia | 0 | 2
  Surgery-wound infection | 0 | 1
  Sweating | 138 | 129
  Syncope | 0 | 3
  Taste disturbance | 1 | 46
  Tearing | 0 | 6
  Thrombocytopenia | 3 | 35
  Thrombosis/embolism | 2 | 5
  Tremor | 0 | 2
  Troponin T (cTnT) increase | 0 | 1
  Urinary frequency/urgency | 86 | 101
  Urinary retention | 13 | 7
  Urinary tr infect w/ neutrop | 0 | 1
  Urinary tr infect w/o neutrop | 1 | 2
  Urinary tr infection, unk ANC | 3 | 2
  Urine color change | 3 | 44
  Urticaria | 3 | 4
  Ventricular arrhythmia | 1 | 0
  Vertigo | 1 | 1
  Vision,NOS | 0 | 1
  Voice change/stridor/larynx | 0 | 6
  Vomiting | 10 | 51
  Weakness (motor neuropathy) | 3 | 6
  Weight gain | 179 | 151
  Weight loss | 12 | 29

4. Secondary Outcome: PSA Progression Free Survival
Description: Measured from date of randomization to date of PSA progression or death due to any cause. PSA progression is defined as a serum PSA level of > 0.2 ng/mL measured on 3 consecutive occasions or in the absence of increasing PSA, a positive bone scan result or other radiographic or histologic evidence of progression will be used. Date of progression will be the date that the first measure of increasing PSA is noted in the series of 3.
Time Frame: Up to 10 Years
Population: Data for trial not collected for analysis.
Arm/Group | Arm I: Bicalutamide + Goserelin | Arm II: Mitoxantrone + Prednisone + Bivalutamid + Goserelin
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: PSA Progression as Surrogate Endpoint for Overall Survival or Disease Free Survival
Time Frame: Up to 10 Years
Population: Data not collected for analysis.
Arm/Group | Arm I: Bicalutamide + Goserelin | Arm II: Mitoxantrone + Prednisone + Bivalutamid + Goserelin
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Arm 1 assessed every 3 months up through 22 months; Arm 2 assessed every 21 days through first four months, and then every 3 months through 22 months
Description: Patients on Arm 1 were monitored for toxicity every 3 months while on hormonal therapy. Patients on Arm 2 were monitored every 21 days while receiving chemotherapy in first 4 months of study, and then every 3 months through hormonal therapy. Patients on either arm maybe have had more frequent monitoring at discretion of the treating physician.
Arm/Group | Arm I: Bicalutamide + Goserelin | Arm II: Mitoxantrone + Prednisone + Bivalutamid + Goserelin
All-Cause Mortality (participants affected / at risk) | 85/469 | 91/460
Serious Adverse Events (participants affected / at risk) | 3/469 | 11/460
Other Adverse Events (participants affected / at risk) | 461/469 | 457/460
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm I: Bicalutamide + Goserelin (N=469) | Arm II: Mitoxantrone + Prednisone + Bivalutamid + Goserelin (N=460)
Reportable adverse event, NOS (General disorders) | 1 | 0
Cardiac ischemia/infarction (Cardiac disorders) | 0 | 1
Thrombosis/embolism (Vascular disorders) | 0 | 1
Flu-like symptoms-other (General disorders) | 1 | 2
Infection with 3-4 neutropenia (Infections and infestations) | 0 | 2
Hyperglycemia (Metabolism and nutrition disorders) | 0 | 1
Pain-other (General disorders) | 0 | 1
Second primary (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 5
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Arm I: Bicalutamide + Goserelin (N=469) | Arm II: Mitoxantrone + Prednisone + Bivalutamid + Goserelin (N=460)
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 6 | 23
Anemia (Blood and lymphatic system disorders) | 71 | 152
Leukopenia (Investigations) | 20 | 319
Lymphopenia (Investigations) | 8 | 51
Neutropenia/granulocytopenia (Investigations) | 13 | 240
Thrombocytopenia (Investigations) | 7 | 36
Edema (Cardiac disorders) | 50 | 65
Hypertension (Cardiac disorders) | 58 | 51
Fatigue/malaise/lethargy (General disorders) | 268 | 365
Rigors/chills (General disorders) | 9 | 24
Sweating (General disorders) | 139 | 133
Weight gain (Investigations) | 186 | 153
Weight loss (Investigations) | 17 | 30
Alopecia (Skin and subcutaneous tissue disorders) | 93 | 133
Dry skin (Skin and subcutaneous tissue disorders) | 17 | 32
Nail changes (Skin and subcutaneous tissue disorders) | 4 | 59
Pruritus (Skin and subcutaneous tissue disorders) | 19 | 27
Rash/desquamation (Skin and subcutaneous tissue disorders) | 59 | 73
Gynecomastia (Endocrine disorders) | 140 | 100
Hot flashes (Endocrine disorders) | 440 | 422
Anorexia (Metabolism and nutrition disorders) | 9 | 44
Constipation/bowel obstruction (Gastrointestinal disorders) | 69 | 133
Diarrhea without colostomy (Gastrointestinal disorders) | 62 | 87
Dyspepsia/heartburn (Gastrointestinal disorders) | 11 | 44
GI-other (Gastrointestinal disorders) | 17 | 25
Nausea (Gastrointestinal disorders) | 31 | 210
Stomatitis/pharyngitis (Gastrointestinal disorders) | 7 | 49
Taste disturbance (Gastrointestinal disorders) | 1 | 46
Vomiting (Gastrointestinal disorders) | 16 | 54
SGOT (AST) increase (Investigations) | 43 | 51
SGPT (ALT) increase (Investigations) | 24 | 33
Hyperglycemia (Metabolism and nutrition disorders) | 61 | 102
Arthritis (Musculoskeletal and connective tissue disorders) | 30 | 32
Joint,muscle,bone-other (Musculoskeletal and connective tissue disorders) | 17 | 34
Muscle weakness (not neuro) (Musculoskeletal and connective tissue disorders) | 58 | 83
Anxiety/agitation (Psychiatric disorders) | 59 | 70
Depression (Psychiatric disorders) | 95 | 99
Dizziness/light headedness (Nervous system disorders) | 42 | 78
Insomnia (Psychiatric disorders) | 93 | 105
Sensory neuropathy (Nervous system disorders) | 59 | 72
Abdominal pain/cramping (Gastrointestinal disorders) | 30 | 53
Arthralgia (Musculoskeletal and connective tissue disorders) | 57 | 77
Bone pain (Musculoskeletal and connective tissue disorders) | 24 | 34
Chest pain,not cardio or pleur (General disorders) | 16 | 23
Headache (Nervous system disorders) | 45 | 88
Myalgia (Musculoskeletal and connective tissue disorders) | 29 | 49
Pain-other (General disorders) | 162 | 173
Cough (Respiratory, thoracic and mediastinal disorders) | 24 | 46
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 35 | 59
Creatinine increase (Investigations) | 10 | 24
Incontinence (Renal and urinary disorders) | 137 | 117
Urinary frequency/urgency (Renal and urinary disorders) | 131 | 130
Urine color change (Renal and urinary disorders) | 4 | 44
Erectile impotence (Reproductive system and breast disorders) | 217 | 171
Libido loss (Reproductive system and breast disorders) | 168 | 134

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-01-15): https://cdn.clinicaltrials.gov/large-docs/24/NCT00004124/Prot_SAP_000.pdf